CLINICAL TRIAL: NCT05199168
Title: Randomized Clinical Trial of Visualization Versus Intraoperative Neuromonitoring of the Recurrent Laryngeal Nerves During Thoracoscopic Esophagectomy
Brief Title: Visualization Versus Intraoperative Neuromonitoring of the Recurrent Laryngeal Nerves During Thoracoscopic Esophagectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E20210023
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-01

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Minimally invasive surgery; Recurrent laryngeal nerves; Intraoperative nerve monitoring
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracoscopic esophagectomy without IONM (No Intervention)
- Thoracoscopic esophagectomy with IONM (Experimental): Intraoperative bilateral recurrent laryngeal nerve monitoring was utilized during dissection of right and left recurrent laryngeal nerve lymph nodes.
  Interventions: Procedure: intraoperative nerve monitoring

INTERVENTIONS:
Procedure: intraoperative nerve monitoring — Intraoperative bilateral recurrent laryngeal nerve monitoring was utilized during dissection of right and left recurrent laryngeal nerve lymph nodes.
  Arms: Thoracoscopic esophagectomy with IONM

SUMMARY:
The clinical value of intraoperative nerve monitoring (IONM) in thoracoscopic esophagectomy remains uncertain. The aim of this randomized clinical trial was to compare the impact of RLN visualization versus IONM on their morbidity following thoracoscopic esophagectomy.

DETAILED DESCRIPTION:
Recurrent laryngeal nerves (RLN) lymph nodes are the most common metastatic areas in esophageal squamous carcinoma. It is a clinical challenge to reduce high incidence of RLN injury rate result from routine dissection of RLN lymph nodes. Thoracoscopic approach may provide a clear operative field and potentially less invasive surgery. But there are still high RLN injury rate only depending on visualization of thoracoscopy. The use of intraoperative nerve monitoring (IONM) was shown very helpful to identify the RLN and associated with a reduction of RLN injury rate in thyroidectomy. However, there is no solid clinical evidence about the effectiveness of utility of IONM in thoracoscopic esophagectomy. Thus, the aim of this randomized clinical trial was to compare the impact of RLN visualization versus IONM on their morbidity following thoracoscopic esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven primary intrathoracic middle and lower esophageal squamous cell carcinoma and will undergo McKeown MIE and bilateral RLN lymph ndoe dissection.
2. No superclavicular lymph node metastasis after preoperative examination.
3. No contraindication for esophagectomy.
4. Expected surgical R0 resection.

Exclusion Criteria:

1. Pre-existed vocal cord dysfunction.
2. Thorax pleural adhesion rendering minimal invasive approach unfeasible.
3. Gastric tube cannot be used for reconstruction.
4. Combined with hemorrhagic disease.
5. Psychiatric patients.
6. Inability to undergo curative resection and/or follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the recurrent laryngeal nerve injury | Till 6 months postoperatively
  The vocal cord function will be assessed by an experienced otolaryngologist using a laryngoscope on 1st postoperative day.RLN palsy will be classified according to the following variables: site (unilateral versus bilateral); duration (temporary [i.e., recovering within 6 months] versus permanent [i.e. not recovering within 6 months])postoperatively.

SECONDARY OUTCOMES:
Number of nodes removed along the right and left RLN | The pathological analysis will be finished within 2 weeks.
  number of lymph node removed
Value of IONM during operation | 1 Day of surgery
Post esophagectomy pneumonia rate | Duration of hospital stay, an expected average of 2~3 weeks.
Operation time (thoracic phase) | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Hongjing Jiang, MD. Ph.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Department of minimally invasive esophageal surgery, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China